CLINICAL TRIAL: NCT07138222
Title: IMmune checkPoint Inhibitor Related gonAdal toxiCiTy in Premenopausal Women and Men With Melanoma
Acronym: IMPACT
Status: Recruiting | Type: Observational
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Other Study IDs: HREC/117978/PMCC; ACTRN12625000395437p (Other: ANZCTR)
Record Dates: First submitted 2025-07-21; First posted 2025-08-22 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-08

CONDITIONS: Melanoma (Skin Cancer)
Keywords: melanoma; skin cancer; immune checkpoint inhibitors; immunotherapy; gonadal toxicity; ovarian function; testicular function; fertility; cytokines; inflammation
MeSH Terms: conditions — Melanoma; Skin Neoplasms; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: premenopausal women with melanoma: Cohort 1: premenopausal women with melanoma, aged ≤45 years, to describe the change in:
  1. ovarian reserve (using serum AMH),
  2. ovarian function (using serum LH, FSH, oestradiol and related sex steroids),
  3. menstrual pattern,
  4. sexual function (using the European Organisation for Research and the Treatment of Cancer questionnaire for the assessment of sexual health in cancer patients (EORTC QLQ SH22), and
  5. circulating cytokine levels before, during and after ICI treatment.
- Cohort 2: men with melanoma: Cohort 2: men with melanoma, aged ≤60 years, to describe the change in:
  6) testicular function (using serum testosterone, FSH, LH, Sex Hormone Binding Globulin (SHBG), inhibin B and related sex steroids), 7) semen parameters (sperm concentration, count, motility, morphology), 8) sexual function (using the EORTC QLQ SH22 questionnaire, International Index of Erectile Function 5 questionnaire (IIEF-5) and the Psychosexual Daily Questionnaire Question 4 (PDQ-Q4)), 9) testicular volume (using orchidometry) in a subset of patients, and 10) circulating cytokine levels before, during and after ICI treatment.

SUMMARY:
This study aims to capture information regarding the effect of immune checkpoint inhibitor (ICI) treatment for melanoma on reproductive organ function and sex hormone levels.

You may be eligible for this study if you are aged 18 years or older, you have been diagnosed with melanoma (Stage II, III or IV) and you are planning to receive ICI treatment. Additional criteria will apply dependent upon your biological sex characteristics.

All participants who choose to enroll in this study will be asked to complete a series of questionnaires and provide blood at 4 of their scheduled treatment visits. These visits are anticipated to add 30 minutes to the scheduled visit time. Male participants will also be asked to provide semen samples at 2 of their scheduled treatment visits. These visits are anticipated to add an additional 30 minutes to the scheduled visit time. No additional or novel treatments will be offered to participants who choose to enroll in this study, this is an observational study only.

It is hoped this research will contribute important information regarding the potential toxic effects of ICI treatment on sexual and reproductive function in patients with melanoma who are receiving ICI treatment.

DETAILED DESCRIPTION:
While immune checkpoint inhibitors (ICIs) are widely used in young melanoma patients and may cause immune-related side effects, their impact on human gonadal function is unknown.

Eligible patients will be identified by their oncologist and provide informed consent. Menstrual/contraceptive history, sexual function questionnaires, and blood samples for gonadal biomarkers will be collected at baseline, 3, 6, and 12 months. Semen and testicular volume (in a subset) will be assessed in men at baseline and 6 months. Patients who cease ICI before the 12 month timepoint will have also have an end of treatment assessment within 4 weeks of stopping treatment.

Patients will be asked to consent to the future use of their biological samples collected during the trial. Samples will be securely stored at Peter MacCallum Cancer Centre, coded, and linked to clinical data. Patients can request sample destruction at any time, but past analyses cannot be undone.

The Sponsor or delegate will manage trial data, while sites are responsible for data entry and resolving queries. Data will be entered into REDCap, a secure system hosted by Peter MacCallum Cancer Centre. Site staff will be trained, and only authorized personnel listed on the delegation log may complete eCRFs.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for inclusion in this trial if all the following criteria apply:

1. Patient has provided written informed consent using the IMPACT Patient Information and Consent form (PICF)
2. Diagnosis of melanoma (Stage II, III or IV) in the de novo or recurrent setting
3. Has a life expectancy of greater than or equal to 1 year
4. Planned to receive ICI treatment, either in the neoadjuvant, adjuvant or metastatic setting, including as:

   * Monotherapy
   * Combination therapy

   For cohort 1: premenopausal women with melanoma
5. Age greater than or equal to 18 and less than or equal to 45 years at the time of signing consent
6. Patient is premenopausal (defined as baseline FSH within the premenopausal range per local laboratory at registration). Women on hormonal contraception who have an abnormal FSH level, will be included if their AMH level is greater than or equal to 1.0 pmol/L at registration
7. AMH level greater than or equal to 1.0 pmol/L at registration

   For Cohort 2: men with melanoma
8. Age greater than or equal to 18 and less than or equal to 60 years at the time of signing consent
9. Fasting morning total testosterone, LH and FSH within the normal range (per local laboratory) at the time registration

Exclusion Criteria:

Patients will not be eligible for inclusion in this trial if any of the following criteria apply:

1. Previous removal of both ovaries (females) or previous removal of both testes or previous vasectomy (males)
2. Planned for or previously had pelvic radiotherapy
3. Any medications within the prior 6 months known to disrupt the hypothalamic pituitary gonadal axis, e.g., GnRH agonists or antagonists, selective estrogen receptor modulators (SERMs), aromatase inhibitors, testosterone, anabolic steroids, etc.
4. Previous or concurrent alkylating or platinum-based chemotherapy within the last 2 years
5. Previous use of ICI
6. History of hypogonadism
7. Presence of any psychological, social, geographical, or other condition for which, in the opinion of the site Investigator, participation would not be in the best interest of the patient (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with melanoma who meet all the inclusion and none of the exclusion criteria will be eligible for the trial.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in ovarian reserve before, during and after ICI treatment | 12 months
  To describe the change in ovarian reserve (using AMH) within 12 months of ICI treatment in premenopausal women with curable melanoma.
Change in testicular function before, during and after ICI treatment | 12 months
  To describe the change in testicular function (using testosterone) within 12 months of ICI treatment in men with curable melanoma.

SECONDARY OUTCOMES:
Change in ovarian function before, during and after ICI treatment | 12 months
  To describe the change in FSH, LH, oestradiol and related sex steroids (DHT, estrone, DHEA, progesterone) by LC-MS assessed on serum within 12 months of ICI treatment in premenopausal women with curable melanoma.
Change in menstrual pattern before, during and after ICI treatment | 12 months
  To describe the change in menstrual pattern (regularity and cycle length) within 12 months of ICI treatment in premenopausal women with curable melanoma.
Change in sexual function before, during and after ICI treatment | 12 months
  To describe the change in sexual function (EORTC SHQ-C22 questionnaire) within 12 months of ICI treatment in premenopausal women with curable melanoma.
Change in circulating cytokine levels before, during and after ICI treatment | 12 months
  To describe the change in circulating cytokine levels (TNF-alpha, IL-1a, IL-1b, IL-10, IL-6, IFN-gamma and granzyme A and B levels) with 12 months of ICI treatment and if cytokine levels are associated with AMH, LH, FSH and oestradiol levels in premenopausal women with curable melanoma.
Change in testicular function before, during and after ICI treatment | 12 months
  To describe the change in testicular function (using serum FSH, LH, Sex Hormone Binding Globulin (SHBG), inhibin B and related sex steroids) within 12 months of ICI treatment in men with curable melanoma.
Change in semen parameters before, during and after ICI treatment | 12 months
  To describe the change in semen parameters within 12 months of ICI treatment in men with curable melanoma.
Change in sexual and erectile function before, during and after ICI treatment | 12 months
  To describe the change in sexual and erectile function (EORTC SHQ-C22 questionnaire) within 12 months of ICI treatment in men with curable melanoma.
Change in testicular volume before, during and after ICI treatment | 12 months
  To describe the change in testicular volume (using orchidometry) in a subset of men with curable melanoma within 12 months of ICI treatment.
Change in circulating cytokines before, during and after ICI treatment | 12 months
  To describe the change in circulating cytokine levels within 12 months of ICI treatment and if cytokine levels are associated with FSH, LH, SHBG, testosterone, and semen analysis in men with curable melanoma.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Wanda Cui, BMEDSCI, MBBS, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (6):
- Australia (6):
  - Melanoma Institute Australia, Sydney, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Cairns Base Hospital, Cairns, Queensland
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Austin Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Australian New Zealand Clinical Trial Registry — https://www.anzctr.org.au/TrialSearch.aspx#&&conditionCode=&dateOfRegistrationFrom=&interventionDescription=&interventionCodeOperator=OR&primarySponsorType=&gender=&distance=&postcode=&pageSize=20&ageGroup=&recruitmentCountryOperator=OR&recruitmentRegion=&ethicsReview=&countryOfRecruitment=&registry=&searchTxt=IMmune+checkPoint+inhibitor+related+gonAdal+toxiCiTy+in+premenopausal+women+and+men+with+melanoma&studyType=&allocationToIntervention=&dateOfRegistrationTo=&recruitmentStatus=&interventionCode=&healthCondition=&healthyVolunteers=&page=1&conditionCategory=&fundingSource=&trialStartDateTo=&trialStartDateFrom=&phase=
- See also: Peter MacCallum Cancer Centre — https://www.petermac.org/research/cohort-studies/impact